CLINICAL TRIAL: NCT02431871
Title: Structural and Functional Sequelae of Developmental Dysplasia of the Hip
Brief Title: Sequelae of Developmental Dysplasia of the Hip
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: EETTMK:94/2014
Record Dates: First submitted 2015-04-20; First posted 2015-05-01 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Developmental Dysplasia of the Hip; Hip Dysplasia
Keywords: Developmental dysplasia of the hip; Hip dysplasia; Occlusal defect
MeSH Terms: conditions — Developmental Dysplasia of the Hip; Hip Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated for DDH in childhood: Subjects have had DDH in childhood. DDH has been diagnosed before age of 1,5 years and treated for.
- Control: Age an sex matched controls of DDH patients

SUMMARY:
The aim of this study is to assess long term effects of developmental dysplasia of the hip (DDH) to overall health and quality of life later in life. We compare hip radiographs, hip symptoms, clinical examination, head asymmetry, dental examination and intraoral scans of 170 children and young adults treated for DDH in their childhood with age and sex matched controls.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip (DDH) is the most common musculoskeletal disorder in infancy. However there are few reports of long term effects of successfully treated DDH. Incidence of DDH in neonatal period is approximately 1-10/1000 depending on screening protocols used, the age of the infant during screening and which ultrasonographic findings are considered normal and which DDH. The prevalence of hip dysplasia in adult population is grossly 4 % when using Wibergs Centre-Edge (CE) ≤ 20° as definition of dysplasia. It is still unclear, what is the relation between adult acetabular dysplasia and developmental dysplasia in children. Hip dysplasia overall is a major contributing factor in hip osteoarthrosis and total hip replacement in young adults.

The aim of this study is to assess long term effects of developmental dysplasia of the hip to overall health and quality of life later in life. We compare hip radiographs, hip symptoms, clinical examination, head asymmetry, dental examination and intraoral scans of 170 children and young adults treated for DDH in their early childhood with age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria for person treated for DDH:

* DDH has been diagnosed by clinical examination, ultrasound examination or by radiological examination and treatment begun before age of 1,5 years.
* Treated in Oulu University Hospital

Exclusion Criteria:

* neurological or developmental condition which can influence hip development such as cerebral palsy or spina bifida
* other significant congenital anomalies of musculoskeletal system such as club feet

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 10-30 years old patientstreated for DDH in early childhood in Oulu University Hospital
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wibergs Centre-Edge Angle | 10 - 30 years after DDH has been treated
  angle degree

SECONDARY OUTCOMES:
The Copenhagen Hip and Groin Outcome Score (HAGOS) | 10 - 30 years after DDH has been treated
  score in numbers
Oral Heath Impact Profile | 10 - 30 years after DDH has been treated
  Oral Heath Impact Profile (OHIP-14) -questionaire to assess Oral Health-related Quality of Life
Occlusal asymmetries | 10 - 30 years after DDH has been treated
  Determined by dental examination and intraoral scan
Presence of facial asymmetry | 10 - 30 years after DDH has been treated
  Determined by 3D -photogrammetric images

OTHER OUTCOMES:
Hip deformity | 10 - 30 years after DDH has been treated
  Determined by hip radiograph
Asymmetry in clinical hip examination | 10 - 30 years after DDH has been treated
  Determined by clinical hip examination

CONTACTS AND LOCATIONS:
Overall Officials: Juhana Leppilahti, Professor, Principal Investigator — University of Oulu; Marita Valkama, Ph.D., M.D, Study Director — University of Oulu, Oulu University Hospital, MRC Oulu; Virpi Harila, Ph.D., Study Director — University of Oulu, MRC Oulu
Locations (1):
- University of Oulu; Oulu University Hospital, Oulu, Finland